CLINICAL TRIAL: NCT06114966
Title: Titanium Versus Soft Metal CAD/CAM Frameworks for All-on-4 Implant Supported Prosthesis. A Study of Peri-implant Changes and Framework Adaptation
Brief Title: Titanium Versus Soft Metal CAD/CAM Frameworks for All-on-4 Implant Supported Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0109023
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Dental Prosthesis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- titanium framework manufactured by dry milling technique (Experimental): All patients will have titanium framework manufactured by dry milling technique and occlusal material made from PMMA FPD
  Interventions: Other: CADCAM
- metal framework manufactured by dry milling/post sintering of Co-Cr soft metal blocks (Experimental): All patients will have metal framework manufactured by dry milling/post sintering of Co-Cr soft metal blocks and occlusal material made from PMMA FPD
  Interventions: Other: CADCAM

INTERVENTIONS:
Other: CADCAM — Milling of Final prosthesis over dental implants using CADCAM milling machine

SUMMARY:
This study is aimed to compare between titanium framework and soft metal framework used for mandibular All-on-4 implant supported prosthesis.

The evaluation will be for:

* Peri-implant soft tissue health including; Plaque index, Probing depth and bleeding index.
* Bone level changes around implant using periapical x-ray after 6 months and 12 months and 18 months from insertion of fixed prosthesis.
* Framework adaptation of titanium framework and soft metal framework using surface matching software.

Patient grouping:

• 20 Patients will be classified into 2 equal groups, first group will receive 4 implants placed according to All on 4 concept supporting screw retained prosthesis with titanium framework manufactured by dry milling technique, second group will receive 4 implants placed according to All on 4 concept supporting screw retained prosthesis with metal framework manufactured by dry milling/post sintering of Co-Cr soft metal blocks.

The evaluation will be for:

• Bone level changes around implant using periapical x-ray after 6 months and 12 months and 18 months from insertion of fixed prosthesis.

DETAILED DESCRIPTION:
This study will compare between titanium framework and soft metal framework used for mandibular All-on-4 implant supported prosthesis regarding bone level changes around implant using periapical x-ray after 6 months and 12 months and 18 months from insertion of fixed prosthesis.

Patient selection Twenty patients will be selected from the out-patient clinic of Prosthodontic Department, Faculty of Dentistry, Mansoura University seeking for prosthetic rehabilitation.

All patients will be informed about all surgical and prosthetic procedures that will be done. Also; they will sign the consent form of ethical committee of faculty of dentistry.

All implants will be installed in the edentulous mandible in each target positions according to their arrangements guided by stereolithographic stent.

* A cone beam computerized tomographic scan will be taken prior to surgery to determine the bone quality and bone volume and construct the surgical stent.
* Infiltration local anesthetic solution will be given for each patient.
* Each patient will receive 2 distally tilted implants in the posterior region anterior to mental foramen followed by 2 anterior implants.
* The stent will allow for optimal positioning, alignment, parallelism, and inclination of the implants for subsequent anchorage and prosthetic support.
* Once implant is placed, multiunit abutment will be placed. Hand tightens will take x-ray to verify seated properly. Torque to 15Ncm for tilted, 35Ncm for straight.
* Antibiotics (Augmentin 1g) will be given 1 hour before surgery and then daily for 5 days. Anti-inflammatory medication will be given after surgery if needed. Analgesics (brufen 600mg) will be given after surgery if needed.
* Immediate loading of the implants will be done by modifying the mandibular denture.
* The mandibular denture will be modified by shortening the flanges and cutting the posterior part till the 1st molar then 3D scanned for recording the correct dimension of each tooth to be concerned during construction of the titanium and soft metal superstructures and the final prosthesis.
* Digital impression technique will be made using intraoral scanner and scan bodies and the resultant scan will be used in construction of titanium and soft metal superstructures with the abutments.

Patient grouping:

* Patients will be classified into 2 equal groups, first group will have titanium framework manufactured by dry milling technique, second group will have metal framework manufactured by dry milling/post sintering of Co-Cr soft metal blocks.
* The fit of the frameworks will be verified intraorally and the final fixed prosthesis will be constructed from PMMA for both groups.

The evaluation will be for:

• Bone level changes around implant using periapical x-ray after 6 months and 12 months and 18 months from insertion of fixed prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous maxillary and mandibular ridges with sufficient mandibular bone height in the inter-foraminal area confirmed with panoramic x-rays.
* All selected patients will be with sufficient inter-arch space and restorative space.
* All selected patients will have apparently healthy ridge covered by compressible oral mucosa and free from any ridge flabbiness.

Exclusion Criteria:

* Patients with systemic diseases that contraindicate implant placement such as hematologic diseases, serious problems of coagulation and diseases of the immune system. Also, metabolic diseases related to bone resorption such as uncontrolled diabetics or osteoporosis will be also excluded
* History of para-functional habits (Bruxism, clenching), smoking and alcoholism.
* History of radiation therapy in the head and neck region.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Peri-implant crestal bone resorption | at time of insertion of prosthesis procedure T(0), 6 months after insertion T(6), 12 months after insertion T(12), 18 months after insertion (T18)
  Crestal bone level will be evaluated by Periapical x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shady, MD, Principal Investigator — Mansoura University Faculty of Dentistry, Prosthodontics department
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No